| 1 | BIG LEAP: A comparison of insulin degludec to continuous subcutaneous infusion of insulir |
|---|---|
| 2 | aspart for basal insulin delivery in type 1 diabetes |
| 3 | Protocol Number: MDEC2018 |
| 4 | INVESTIGATOR INITIATED STUDY PROPOSAL |
| 5 | Universal Trial Number: U1111-1199-8692 |
| 6 | Mountain Diabetes and Endocrine Center |
| 7 | 1998 Hendersonville Rd, Bldg 31 |
| 8 | Asheville, NC, USA |
| 9 | |
| 10 | Correspondence to: |
| 11 | Wendy Lane MD |
| 12 | Director of Clinical Research |
| 13 | Mountain Diabetes and Endocrine Center |
| 14 | Phone: (828) 684- 9588 |
| 15 | Cell: (828) 778-5006 |
| 16 | Fax: (828) 684-9626 |
| 17 | Email: mountaindiabetes@msncom |

### **BACKGROUND AND SIGNIFICANCE**

18 19

20

2122

23

24

25

26

27

28 29

30 31

32

33

34

35 36

37

38

39

Physiologic insulin replacement for the treatment of type 1 diabetes, or intensive insulin therapy, is administered either by multiple daily injections (MDI) of insulin or via continuous subcutaneous insulin infusion (CSII) via insulin pump. Since its inception in the 1970's, CSII has improved continuously in terms of both the devices and the rapid acting insulin analogues they deliver so that today's insulin pumps are considered the "gold standard" of intensive insulin therapy. However, CSII has only shown advantages over MDI regimens which used older basal insulin products including intermediate-acting insulin (NPH) and first generation insulin analogues (glargine and detemir) including reducing the incidence of hypoglycemia, improving overall glycemic control and improving glycemic variability (1,2). CSII also has advantages in terms of patient convenience and comfort by eliminating the need for multiple daily insulin injections, portability of insulin, and the use of computerized bolus calculators to assist with bolus calculations. However, patients treated with CSII continue to show significant glycemic variability owing to different absorption characteristics of insulin infused subcutaneously at different body sites and due to the inherent variability of absorption of rapid-acting insulin analogues even when infused continuously in sub-unit quantities for basal insulin delivery by modern insulin pumps.

Insulin degludec is a new ultralong-acting insulin analogue with a unique mechanism of protraction giving it a flat, peakless pharmacodynamic profile with a coefficient of variation of the glucose infusion rate of approximately 25% that of insulin glargine in glucose clamp studies

40 and a half-life of 25 hours (3). Insulin degludec has also been shown to have a reduced incidence of hypoglycemia compared to insulin glargine in a head-to head clinical trial in 41 patients with type 1 diabetes. (4). Whether insulin degludec might provide equivalent basal 42 insulin coverage with a flatter 24 hour glycemic profile compared to CSII using a rapid-acting 43 44 insulin analogue is currently not known as these have not been compared in a clinical trial. Part 45 of the reason for this is because patients using CSII use a pump for both the basal and bolus component of their insulin regimen; currently, no "bolus only" insulin delivery device exists. 46 Also, there was no compelling reason until now to study a hybrid model for basal/bolus insulin 47 48 regimens since there was no true 24 hour basal insulin product which had any therapeutic advantage over basal insulin delivered by CSII. Furthermore, it is now recognized that the use 49 50 of insulin infusion sets of various design in CSII lead to increased glucose variability by virtue of local inflammation and micro-occlusions of the sets, which interfere with consistent insulin 51 52 basal delivery (5). Insulin degludec, however, appears in clinical use to possibly have a flatter 53 glycemic profile than CSII can provide, with equivalent or even lower glycemic variability and 54 less hypoglycemia. If so, patients with type 1 diabetes may achieve better overall glycemic 55 control with, and therefore prefer, a daily injection of insulin degludec for their basal insulin 56 needs in combination with their pump (with its bolus calculator) for their bolus insulin needs.

57 The purpose of this investigator-initiated trial is to compare the effect of a daily injection of

insulin degludec vs. basal insulin delivery via CSII, both in combination with bolus insulin 58

59 delivery via the patient's usual insulin pump with insulin aspart, on glycemic variability, overall

60 blood glucose control and incidence of hypoglycemia, all assessed by continuous glucose

monitor (CGM), as well as patient satisfaction, in patients with type 1 diabetes currently using 61

62 CSII.

63

75

76

### **SPECIFIC OBJECTIVES**

64 The primary objective of this trial is to determine whether insulin degludec will provide an

equally stable and consistent basal glycemic profile with lower glycemic variability as 65

determined by CGM compared to insulin aspart delivered by CSII in patients with type 1 66

diabetes experienced in use of insulin pump therapy. Specifically, this study will determine if 67

the percent time in the target glycemic range (70 to 180 mg/dl) by CGM is superior using insulin 68

69 degludec than continuously infused insulin aspart, and if degludec is associated with lower GV

70 as assessed by the standard deviation (SD) of the mean daily glucose by CGM. Particular

attention will be given to the nocturnal glucose profile (from midnight to 6 am) which most 71

72 closely reflects basal insulin action as it is typically the time of day least affected by bolus

73 insulin, food intake or exercise. Quality of life questionnaires regarding treatment preference

74 will be used to capture patient preference for method of basal insulin delivery.

### **RESEARCH DESIGN AND METHODS**

# Study hypothesis

It is anticipated, based on the low glycemic variability of insulin degludec shown in glucose clamp studies and seen in clinical practice, that insulin degludec will provide more stable 24 hour basal insulin action than insulin aspart by CSII in patients with type 1 diabetes.

# **OUTCOME MEASURES/SPECIFIC ENDPOINTS**

## **Primary endpoint**

Percent time in euglycemia (BG 70 to 180 mg/dl) by CGM during the final 14 days of each treatment period during steady state (with basal insulin delivery as either one daily injection of insulin degludec or as insulin aspart via CSII).

## **Key secondary endpoints**

- 1. SD of interstitial fluid glucose by CGM for 2 week period during each basal insulin delivery method. (Note: because the Dexcom Platinum G5 CGM is currently only FDA approved for 7 days of use, two contiguous CGM periods using 2 sensors, each for 7 days, will be performed to capture 2 weeks of continuous CGM data.) Dexcom G6 is approved by FDA for 10 days of use so 2 sensors will be used during the CGM periods.
- 2. SD of blood glucose by CGM during the nocturnal period (midnight to 6 am) during each basal insulin delivery method

# Other secondary endpoints

- 1. Percent time in hypoglycemia by CGM, captured at 2 levels of hypoglycemia: BG ≤ 54 mg/dl (level 2) and BG 55-69 mg/dl (level 1), for each basal insulin treatment.
- 2. Percent time in normoglycemia (BG 70 to 140 mg/dl) by CGM during each basal treatment period.
- 3. Time to recovery from level 2 hypoglycemia (BG >70 with resolution of symptoms) on each treatment. If a second event (BG < 70 mg/dl) occurs within 60 minutes of a previous hypoglycemic event, this will be considered part of the same hypoglycemic episode.
- 4. Patient satisfaction by TRIM-D and TRIM-DD questionnaires with each basal insulin treatment.
- 5. HbA1c after 20 weeks of each basal insulin treatment.
- 6. Total daily insulin dose, total basal insulin dose, and total bolus insulin dose on each treatment.

- See Table 1: Study Visit Table for study procedures at each visit and when specific endpoints will be measured.
  - STUDY TYPE

- 115 This will be a randomized, cross-over, open label, single-center study consisting of a 20 week
- period on each of two basal insulin delivery methods, both in combination with insulin aspart
- with boluses taken by insulin pump. Each 20 week period will consist of a 4 week insulin
- optimization period for titration of basal and bolus insulin doses, followed by a 16 week
- maintenance period. The final 2 weeks of the maintenance period during each treatment arm
- will be used for endpoint data collection. The treatment sequence will occur in random order.
- 121 The study population will include patients with type 1 diabetes with good baseline glycemic
- control who are experienced in the use of both CSII and CGM; the cross-over design allows each
- subject to serve as his or her own control.

# STUDY POPULATION

- 125 In order to confirm a 10% improvement in the time spent in euglycemia by CGM with 85%
- power, 47 subjects will be studied. Thus, between 55 and 60 subjects will be screened to allow
- for a 10% drop-out rate. (See "Statistical Analysis Plan" for sample size calculation.)

### 128 INCLUSION CRITERIA

- 129 1. Male and female patients > 18 years of age with type 1 diabetes using CSII with any pump for
- 130 > 12 months.

124

- 2. Females must be using adequate contraception, defined as oral contraceptive pill, barrier
- method of contraception, or surgical method (tubal ligation or hysterectomy).
- 133 3. Good glycemic control (HbA1c  $\leq$  8.0%).
- 4. Patients are experienced in carbohydrate counting, evidenced by pump downloads showing
- frequent meal boluses with realistic carbohydrate entries, few over-rides of the pump bolus
- calculator, few to no omitted boluses (at least 3 boluses per day), and post-meal glucose levels
- generally below 200 mg/dl indicating accurate carbohydrate assessment.
- 138 5. Patients are regular (>85% of time) users of the Dexcom G5 or G6 CGM.
- 6. Pump download confirms correct use of insulin pump features, including appropriate use of
- bolus calculator with minimal overrides, entering carbohydrate content of meals, at least 3
- boluses taken per day, appropriate use of correction boluses, and infusion set changes every 2
- 142 to 3 days.

150 151

152

- 7. No serious comorbidities including: retinopathy requiring active intervention, eGFR < 30, CV
- event within the previous 6 months, active malignancy with ongoing treatment, any condition
- requiring chronic use of systemic glucocorticoids, or any other condition which in the opinion of
- the investigator would interfere with the subject's ability to comply with the study protocol or
- 147 acutely affect insulin requirements.
- 148 8. Able to comply with study protocol.
- 9. Ability to provide written informed consent prior to any study-related procedures.

## **EXCLUSION CRITERIA**

- 1. Subjects with type 2 diabetes.
- 154 2. Subjects with HbA1c > 8.0%

- Subjects not using CSII and CGM (ie, on MDI)
  - 4. Subjects inexperienced in the use of CSII, or whose pump download shows poor utilization of bolus calculator features, ie fewer than 2 boluses per day, lack of correction boluses, frequent overrides of the recommended boluses, unrealistic carbohydrate entries (suggestive of under-bolusing), not changing infusion set at least every 3 days, or other evidence of poor insulin pump usage.
  - 5. Subjects inexperienced in or not regular users (>85% of time) of Dexcom G5 or G6 CGM
  - 6. Subjects who are using a Medtronic pump with low blood glucose suspend who are unwilling to use the Dexcom CGM or to disengage the low blood glucose suspend feature of the pump.
  - 7. Use of any other CGM than Dexcom G5 or G6.
  - 8. Serious concomitant illness.
  - 9. Females unwilling to use adequate contraception, intending to become pregnant, or breastfeeding.
  - 10. Known or suspected allergy to study products, their excipients or related products.
  - 11. Previous participation in this trial. Note: subjects who screen fail because of A1c may rescreen once if, in the opinion of the investigator, the HbA1c was explainable (ie, recent steroid injection or illness, etc) and atypical for the subject.
  - 12. Hypoglycemic unawareness.
  - 13. Episode of severe hypoglycemia (requiring assistance for treatment) within the previous 90 days.

### 177 WITHDRAWAL CRITERIA

- 178 Subjects may withdraw at will for any reason.
- 179 Females who become pregnant will be discontinued from the study.
- Subjects who do not comply with CGM use or switch from use of CSII to MDI will be discontinued.

Subjects who are discontinued from the study will not be replaced.

## **RATIONALE FOR THE STUDY POPULATION**

A population of well controlled patients with type 1 diabetes who are experienced in the use of both CSII and CGM was chosen in order to assess the effect of the change in glycemic profile using two different methods of basal insulin delivery. Studying a population with expertise in diabetes self-management with these devices will minimize the effect of incorrect device use and allow assessment of the effect of the change of insulin regimen itself. Allowing the subjects to use their insulin pumps for bolus insulin delivery, as they are accustomed, will minimize the chances of skipping meal boluses and correction doses.

Replacing basal insulin delivery by CSII with a single daily injection of degludec will add minimal, if any, treatment burden which will be offset by potential therapeutic benefits. These benefits include the potential for reduced glycemic variability and the elimination of the risk of

hyperglycemia and DKA with basal insulin interruption which can occur with infusion set occlusion or dislodgement inherent to CSII. Subjects may also enjoy the freedom afforded by a basal insulin injection which will allow them to disconnect from their pumps safely without sacrificing glycemic control for prolonged periods of time (which is not an option using CSII for basal insulin delivery).

#### **VISIT PROCEDURES**

Please see pages 16-18 for "Visit Procedures", which describes a detailed list of procedures and assessments at each visit, and page 19 for the "Study Flow Sheet", which summarizes study-related procedures at each visit in spreadsheet format.

#### ASSESSMENTS OF EFFICACY

## **Primary endpoint**

Percent time spent in euglycemia by CGM: data will be downloaded from the Dexcom G5 or G6 (either by download of receiver or from Dexcom Clarity cloud-based application); this will yield the percent time in euglycemia, hyperglycemia, hypoglycemia and SD for endpoint analyses.

# Other endpoints

1. HbA1c: This will be measured by central laboratory (LabCorp, Burlington, NC). 2. GlycoMark (1,5 anhydroglucitol) will be measured by commercial assay (LabCorp, Burlington, NC). All laboratory specimens will be drawn and processed by site staff and shipped under required conditions to LabCorp by courier with pick-up daily. GlycoMark is a marker of glycemic variability which essentially reflects postprandial glucose control. It will be captured as a safety measure to ensure that change of method of basal insulin delivery does not impact postprandial glucose control in any way, since patients using CSII may on occasion have increased postmeal basal insulin infusion rates (to compensate for inadequate mealtime insulin dosing) which cannot be reproduced in the degludec treatment arm.

### **ASSESSMENTS OF SAFETY:**

Hypoglycemia will be captured by fingerstick BG and by CGM. All episodes of severe hypoglycemia (requiring assistance) will be documented and reported as AE's in diaries. Categories of hypoglycemia that will be captured include: percent time in two categories of hypoglycemia (BG < 54 mg dl and 55-69 mg/dl) by CGM, episodes of symptomatic BG-confirmed hypoglycemia (<54 mg/dl), nocturnal hypoglycemia and severe hypoglycemia. In the event where the SMBG and the CGM readings are discordant, the SMBG will be considered the primary source.

Time to recovery from hypoglycemia, defined as BG  $\geq$  70 with resolution of symptoms, during each treatment will also be captured.

#### OTHER ASSESSMENTS

242243244

Patient satisfaction with each study treatment will be assessed by TRIM-D and TRIM-DD questionnaires.

245246247

#### ASSESSMENT OF SUBJECT COMPLIANCE

248249

250

251

252

Compliance of study subjects with use of CSII and CGM will be assessed by review of device downloads which capture percent time devices are used, set changes, boluses and carbohydrate intake. Since subjects will be using their insulin pumps to bolus, all bolus insulin doses and carbohydrate intake will be captured in both treatment arms by review of insulin pump downloads at each study visit.

253254255

256

257

Compliance with administration of basal insulin during the degludec treatment arm will be assessed by documentation of insulin doses and times in subject diaries. Number of missed injections will be captured during the degludec treatment arm; number of infusion set changes, set occlusions, and missed boluses will be captured during both treatment arms.

258259260

## STATISTICAL CONSIDERATIONS

261262

# **Sample Size Determination**

263

264

265266

267268

The subjects in a recent study (4) should closely reflect the population we are going to study. Using the statistics from that source as an estimate of population parameters, power analyses were done for: (1) percent time in euglycemia (BG 70 to 180 mg/dl), desired effect size 0.4, (2) SD of BG by CGM, desired effect size 0.44, and (3) HbA1c, desired effect size 0.44. The repeated independent variable is degludec vs CSII. These a priori analyses – using G\*Power, version 3.1.9.2 <a href="http://www.gpower.hhu.de/en.html">http://www.gpower.hhu.de/en.html</a> – assumed a Type I error of .05 and a power of .85

The sample size estimate required for percent time in euglycemia was the largest at n = 47.

269270

271

272 Allowing for a 10% dropout rate a final sample size of 53 will be sought – more if possible.

273

# **Statistical Methods**

(Type II error of .15).

274275276

Ho: For Type 1 DM subjects using degludec vs CSII, there is no difference between mean percent time in euglycemia, mean SD of BG by CGM, or mean HbA1c.

277278279

Ha: For Type 1 DM patients using degludec vs CSII, there will be mean differences between percent time in euglycemia, SD of BG by CGM, and HbA1c. (No one tailed tests are planned.)

280 281 282

# **Dependent Variable**

One group of patients will first use degludec for 20 weeks then switch to CSII for 20 weeks. As all eligible patients who sign the IRB consent form are identified, a random number will be

generated to determine the treatment with which they begin first. The other group of patients will start with CSII and after 20 weeks switch to Tresiba for 20 weeks. Randomization sequence will be determined by computerized randomization program. All patients will receive both treatments unless they drop out. Dropouts are unlikely since the participants are all regular continuing patients of the site's clinical practice.

290

- Since each patient will be measured twice insulin degludec vs CSII by pump this repeated measure will be the dependent variable.
- Since study participants are all ongoing patients of the three physicians at the site, there should be no missing data, per-protocol, or intention-to-treat issues. Only patients who complete the entire 46-week study will be used in the final analysis.

296297

No continuous or ratio variables will be categorized.

298

299 No interim analysis will be performed.

300

301

### Control/covariate variables

- These will be recorded at the beginning of the study to help reduce error variance in the
- 303 dependent measures:
- 1) Time elapsed since diagnosis of Type 1 DM (ratio variable)
- 305 2) Age (ratio variable)
- 3) Physician attending each patient there are 3 physicians (nominal).
- 307 4) Whether each patient started with CSII by pump or insulin degludec (nominal)
- 308 5) Race of patient (if there is any variability; unlikely) (nominal).

309 310

317

# Statistical Analysis

- 311 Statistical analyses will be performed using STATA version 15.0, revision 25, released
- 312 September 2017. (www.stata.com)
- 313 Since all the dependent variables are interval and the independent and control/covariate
- variables are a mixture of ratio and nominal, a General Linear Model for Repeated Measures
- analysis can be used. Depending on the final sample sizes a hierarchical stepwise analysis could
- be performed to identify the more useful control/covariate variables.

#### DATA HANDLING AND RECORD KEEPING

- The study data (CGM data and laboratory endpoints including HbA1c and GlycoMark) will be
- 319 uploaded and stored in the cloud in HIPAA-compliant electronic files. Pertinent data for
- endpoint safety and efficacy analyses will be entered into and electronically filed in password-
- 321 protected Excel spreadsheets. Hypoglycemia diaries will be on paper and stored as source
- documents along with paper CRF's capturing study-related procedures (history, physical exam,

| 323<br>324 | vital signs, con meds, AE's) at each visit. Patients will complete TRIM-D and TRIM-DD questionnaires, and responses will be tabulated into Excel spreadsheets for statistical analysis. |
|---|---|
| 325<br>326 | All paper source documents and CRFs will be stored on site. All electronic data will be stored in the cloud in HIPAA-compliant electronic files. |
| 327 | ETHICAL CONSIDERATIONS |
| 328<br>329<br>330 | The sponsor (Mountain Diabetes and Endocrine Center), its investigators and site staff will comply with all applicable regulatory and legal requirements, ICH GCP guidelines and the Declaration of Helsinki in obtaining and documenting the informed consent. |
| 331<br>332<br>333<br>334<br>335<br>336<br>337 | Informed consent will be obtained by a medically qualified site member (MD or RN) after each subject has had time to review the informed consent document and have any questions about the study answered. This is performed in a conference room at the study site in a private and unhurried fashion. The subjects may bring family members with them to witness the informed consent process. The informed consent documents will be paper documents that will be retained at the site, signed by the subject and investigator, and a copy will be provided to each subject. |
| 338<br>339<br>340<br>341 | Upon approval of the study protocol, the study will be submitted for approval to IntegReview IRB in Austin, Texas for review and approval. The informed consent document will include information about the IRB and contact information for the IRB, the site, and the study principal investigator. |
| 342<br>343 | The study will be conducted in accordance with ICH GCP guidelines and the Declaration of Helsinki. |
| 344 | STUDY SCHEDULE |
| 345 | Planned recruitment period: 6 to 9 months |
| 346 | Expected milestones: Start of study: immediately upon IRB approval (March 2018) |
| 347<br>348 | First patient first visit (FPFV): within 1 week of IRB approval (site is ready to begin recruitment with subjects available to start upon protocol and IRB approval and obtaining study insulin) |
| 349 | Last patient first visit (LPFV): within 6 to 9 months of FPFV |
| 350 | Last patient last visit: 46 weeks after LPFV |
| 351 | Estimated study duration (FPFV to LPLV): 14 months (March 2018 to May 2019) |
| 352 | Completion of final study report: within 6 weeks of study completion |
| 353 | Time to submission of study for publication: within 12 weeks of study completion |
| 354 | STUDY DRUGS AND MATERIALS |

- 355 Study medication: insulin degludec (Tresiba) U100 or insulin degludec (Tresiba) U200 (Novo
- Nordisk) with insulin aspart (administered as bolus insulin via insulin pump) (Novolog, Novo
- Nordisk) for one treatment arm; insulin aspart (Novolog) administered by CSII for both basal
- 358 and bolus insulin in second treatment arm.
- 359 Study Devices: subjects' own insulin pumps will include Medtronic (530, 730 models; no low
- 360 blood glucose suspend models or closed loop pumps will be used), Animas Ping, Animas Vibe,
- 361 Tandem T-slim and Insulet Omnipod.

363

371

383

The study CGM will be Dexcom G5 or G6.

## PACKAGING AND LABELLING OF STUDY MEDICATION AND DEVICES

- 364 Study insulins (insulin degludec and aspart) will be distributed at study visits to each subject
- 365 from the site. Insulin degludec will be supplied in injection pens (5 per box for U100 and 3 per
- box for U200). Insulin aspart will be supplied in vials (as bolus insulin will be administered via
- insulin pump.) Subjects will use their own insulin pumps and pump supplies during the study.
- Dexcom sensors will be supplied for a two week period (using one sensor weekly) at baseline
- and for the final two weeks of each treatment period. These will be distributed and placed at
- 370 CGM dispensing/insertion site visits (see study visit flow sheet).

### STORAGE AND DRUG ACCOUNTABILITY OF STUDY MEDICATION

- 372 Study insulins will be received in temperature-controlled containers and the temperature of the
- 373 medication upon receipt will be recorded. Study insulins will be stored at the study site in
- 374 refrigerators maintained between 2 and 8 degrees Celsius; the temperature will be monitored
- and recorded daily. No trial medication will be dispensed to any individual not enrolled in the
- 376 study. All medication used in the study will be recorded in the CRF at each study dispensing
- visit. Subjects will be provided with sufficient study insulin for study completion.
- 378 Subjects will be instructed not to refrigerate opened insulin degludec (Tresiba U100 & U200)
- and to store the product at room temperature. Properly stored opened insulin degludec can be
- used for up to 8 weeks (7). Subjects may choose to refrigerate or not refrigerate an opened vial
- of insulin aspart (Novolog), maintaining the vial at a temperature of less than 86°F (30°C) for up
- 382 to 4 weeks (8).

### **AUXILIARY SUPPLY**

- 384 Study subjects will use their own insulin pumps and insulin pump supplies.
- 385 Dexcom glucose sensors (6 per subject) will be purchased by the site and supplied to subjects
- for two weeks at 3 times (baseline and for the final two weeks of each treatment period).
- 387 Subjects will use their own CGM receiver devices which will be downloaded at appropriate
- 388 study visits. Site will have back up receivers to supply to subjects in case of loss or malfunction
- of subject's own device (not likely). Subjects will use their own sensors for each treatment
- 390 period except for the 3 two week periods of CGM data capture as described above.

| 391 | |
|---|---|
| 392 | |
| 393 | RANDOMIZATION AND BLINDING |
| 394<br>395<br>396 | This is an unblinded study as the two basal insulin delivery methods (degludec via injection vs. aspart via CSII) cannot be blinded. For a description of the randomization and treatment allocation, please refer to the Statistical Methods section above. |
| 397 | CONCOMITANT ILLNESSES AND MEDICATIONS |
| 398<br>399<br>400<br>401<br>402<br>403<br>404<br>405<br>406<br>407<br>408 | Definitions: Concomitant illness: any illness that is present at the start of the trial (at the first study visit). Concomitant medication: any medication other than the trial product(s) that is taken during the trial, including the screening and run-in periods. Details of all concomitant illnesses and medication will be recorded at trial entry (at the first study visit). Any changes in concomitant medication will be recorded at each visit. The information collected for each concomitant medication will include start date, stop date or continuing, and indication. For each concomitant illness, date of onset, date of resolution or continuing, will be recorded. ADVERSE EVENTS |
| 409<br>410<br>411<br>412<br>413<br>414 | Adverse events will be captured at each study visit and recorded on CRF's. Special AE and SAE reporting forms have been created to capture these events. SAE's will be reported within 24 hours of discovery to appropriate local and federal authorities as well as to the IRB when appropriate. The study site will comply with all local legal, regulatory, and IntegReview IRB requirements. |
| 415<br>416<br>417<br>418<br>419 | Mountain Diabetes and Endocrine Center, its investigators, and site staff will be responsible for reporting of all adverse events including serious adverse events (SAE), suspected unexpected serious adverse reactions (SUSARs) and serious adverse drug reactions (SADRs) to the competent authority and independent ethics committee/institutional review board based upor federal regulations and local/IRB policies. |
| 420<br>421<br>422<br>423 | Mountain Diabetes and Endocrine Center, its investigators, and site staff will report to Novo Nordisk all SAEs, SUSARs, and SADRs at the same time such events are reported to regulatory authorities or within 15 days from the site becoming aware of such adverse events, whichever comes first. |
| 424<br>425 | Mountain Diabetes and Endocrine Center, its investigators, and site staff will collect the following information at minimum for each of these events: |
| 426<br>427 | 1. Study name |

- 428 3. Event (with appropriate diagnosis)
- 429 4. Drug
- 430 5. Reporter identification
- 431 Also 6) Causality, and 7) Outcome might be reported, if appropriate.

#### 432 **DEFINITIONS**

### 433 Adverse Event (AE):

- 434 An AE is any undesirable medical event occurring to a subject in a clinical trial, whether or not
- related to the trial product(s). This includes events reported from the first trial related activity
- after the subject has signed the informed consent and until post treatment follow-up period as
- defined in the protocol. This will also include any events related to the malfunction of a
- 438 medical device (i.e. an insulin pump or Dexcom CGM). The following will not be recorded as
- 439 AEs, if recorded as medical history/concomitant illness on the CRF at screening:
- Pre-planned procedure, unless the condition for which the procedure was planned has

  \*\*The planned from the first trial related estimits of the procedure was planned the informed corner.
- worsened from the first trial related activity after the subject has signed the informed consent
- Pre-existing conditions found as a result of screening procedures

# Clinical Laboratory Adverse Event:

- 444 A clinical laboratory AE is any clinical laboratory abnormality regarded as clinically significant,
- i.e. an abnormality that suggests a disease and/or organ toxicity and is of a severity which
- requires active management, (i.e. change of dose, discontinuation of trial product, more
- 447 frequent follow-up or diagnostic investigation).

# 448 449

443

### Serious Adverse Event (SAE):

- 450 A serious AE is an event that results in any of the following:
- 451 Death
- A life-threatening\* experience
- In-patient hospitalization or prolongation of existing hospitalization
- 454
   A persistent or significant disability/incapacity
- 455 A congenital anomaly/birth defect
- Important medical events that may not result in death, be life-threatening\*, or require
   hospitalization may be considered an SAE when, based upon appropriate medical judgement,
   they may jeopardise the subject and may require medical or surgical intervention to prevent
   one of the outcomes listed in this definition. Suspicion of transmission of infectious agents
- 460 must always be considered an SAE.
- \*The term life-threatening in the definition of SAE refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it was more severe.

# 464 465

# **Suspected Unexpected Serious Adverse Event (SUSAR):**

- 466 Mountain Diabetes and Endocrine Center will inform the appropriate regulatory authorities, the
- 467 IRB, and Novo Nordisk of trial product-related SUSARs in accordance with reporting
- 468 requirements and GCP guidelines.

469 470 **Serious Adverse Drug Reaction (SADR):** 471 An adverse drug reaction (ADR) is an adverse event for which a causal relationship 472 (Possible/Probable relation) between the study drug and the occurrence of the event is suspected. The ADR will be classified as serious if it meets one or more of the seriousness 473 474 criteria. 475 Medical Events of Special Interest (MESI): A MESI is (1) a medication error (e.g. wrong drug 476 477 administration or wrong route of administration) or (2) a suspected transmission of an 478 infectious agent via the product 479 480 **Non-Serious Adverse Event:** A non-serious AE is any AE which does not fulfill the definition of an SAE. 481 482 483 **Severity Assessment Definitions:** • Mild: Transient symptoms, no interference with the subject's daily activities 484 485 Moderate: Marked symptoms, moderate interference with the subject's daily activities 486 Severe: Considerable interference with the subject's daily activities, unacceptable 487 488 Relationship to study medication Assessment Definitions: 489 Probable: Good reason and sufficient documentation to assume a causal relationship 490 • Possible: A causal relationship is conceivable and cannot be dismissed 491 Unlikely: The event is most likely related to an etiology other than the trial product 492 **Outcome Categories and Definitions:** 493 494 495 • Recovered: Fully recovered or by medical or surgical treatment the condition has returned to 496 the level observed at the first trial related activity after the subject signed the informed 497 consent 498 • Recovering: The condition is improving and the subject is expected to recover from the event. This term should only be used when the subject has completed the trial 499 500 Recovered with sequelae: As a result of the AE, the subject suffered persistent and significant disability/incapacity (e.g. became blind, deaf, paralysed). Any AE recovered with 501 sequelae will be rated as an SAE 502 503 Not recovered Fatal 504 505 Unknown 506 507 Collection, Recording, Evaluating, and Reporting of Adverse Events 508

509 510

511

All events meeting the definition of an adverse event will be collected, reported, and evaluated

from the first trial-related activity after the subject has signed the informed consent and until

the end of the post-treatment follow-up period as stated in the protocol. All adverse events

resulting from incorrect storage or usage of study product as per product labelling, if applicable, will be reported to the appropriate institutions (7,8). The investigator will copy Novo Nordisk when expediting SAE information to health authorities and will report all SAEs related to Novo Nordisk products to the local Novo Nordisk affiliate safety department. SAE submission to Novo Nordisk will be within 15 days from the investigator's first awareness of the event.

## Follow-up of Adverse Events

During and following a subject's participation in this clinical trial, Mountain Diabetes and Endocrine Center, its investigators and site staff, will provide adequate medical care to the study subject for any study-related adverse events, including clinically significant laboratory values related to the study. This medical care for study subjects will be provided regardless of their insurance status.

All adverse events classified as serious or severe or possibly/probably related to the trial product will be followed until the subject has recovered and all queries have been resolved. For cases of chronic conditions, follow-up until the outcome category is "recovered" is not required, as these cases can be closed with an outcome of "recovering" or "not recovered". All other adverse events will be followed until the outcome of the event is "recovering" (for chronic conditions), or "recovered" or until the end of the post-treatment follow-up stated in the protocol, whichever comes first, and until all queries related to these AEs have been resolved.

# **Pregnancy**

Study subjects will be instructed to notify the site and study physician immediately if they become pregnant.

Mountain Diabetes and Endocrine Center, its investigators and site staff, will report to Novo Nordisk any pregnancy occurring during the trial period. Reporting of pregnancy by the site will occur within the same timelines described above for reporting of Adverse Events.

Pregnancy complications will be recorded as adverse event(s). If the infant has a congenital anomaly/birth defect this must be reported and followed up as a serious adverse event.

# **Precautions/Insulin Over-dosage**

547 Study subjects will be prescribed glucagon kits and treatment of hypoglycemia will be reviewed 548 with subjects upon enrolment into the study.

# **LIABILITY AND SUBJECT INSURANCE:**

During and following a subject's participation in trial, Mountain Diabetes and Endocrine

Center and the study physicians will provide adequate medical care to the study subject for

any study-related adverse events, including clinically significant laboratory values related to

the study. This medical care for study subjects will be provided regardless of their insurance status.

Mountain Diabetes and Endocrine Center and its investigators will be responsible for the conduct of the study and agree to defend, indemnify, and hold harmless Novo Nordisk, any of its parent companies, affiliates, or subsidiaries, and their respective officers, directors, employees, agents, representatives, distributors, salespersons, customers, licensees, and end-users from and against any claim, suit, demand, loss, damage, expense or liability imposed by any third party arising from or related to: (a) any breach of sponsor-investigator's obligations or representations; or (b) sponsor-investigator's negligent or grossly negligent use or willful misuse of the study drug, the results, or services derived therefrom. This indemnification shall not apply in the event and to the extent that a court of competent jurisdiction or a duly appointed arbiter determines that such losses or liability arose as a result of Novo Nordisk's gross negligence, intentional misconduct, or material breach of its responsibilities.

### **EVALUABILITY OF SUBJECTS**

Only the principal investigator has the authority to exclude any subjects or data observations after the initiation of the study, initial selection of subjects, and beginning of data collection. Possible reasons for such actions might be (1) questionable validity or reliability of data collection or measurement techniques for a particular subject, (2) misrepresentation of initial selection criteria by a subject, or (3) changes in the health conditions of subjects that might affect the reliability or validity of measurements or accuracy of data collection procedures. The reasons for any such action will be carefully documented by the principal investigator and kept on file for the actionable subject.

#### PREMATURE TERMINATION OF STUDY

The study will only be discontinued prematurely in the unlikely event of an unforeseen safety concern arising from the study protocol.

## **PUBLICATION PLAN**

Upon approval, the study will be registered with www.clinicaltrials.gov.

Upon study completion, the study results will be submitted in a manuscript to a peer-reviewed journal. It is anticipated that the study results will be of sufficient interest and importance to be presented at one or more national meetings, notably ADA, AACE and AADE.

### REFERENCES

1. Miller KM et al. Diabetes Care 2015; 38: 971-978

- 595 2. Misso ML et al. Cochrane Database Syst Rev. 2010(1):CD005103
  - 3. Heise T et al. Diabetes Obes Metab 2012 Sep;14(9) 859-64
  - 4. Lane W et al. JAMA. 2017; 318 (1): 33-44

- 5. Hauzenber JR et al. *Diab Technol Therapeutics* 2017 http://online.liebertpub.com/doi/full/10.1089/DIA.2017.0175
- 6. Bergenstal R et al. JAMA. 2016; 316(13):1407-1408
- 7. Novo Nordisk. (2015). TRESIBA® (insulin degludec injection) Label. 28-29
- 8. Novo Nordisk. (2000). NovoLog (insulin aspart [rDNA origin]) injection label. 21-22

### APPENDIX: METHOD OF CONVERSION OF BASAL INSULIN BY CSII TO DEGLUDEC

Upon randomization to insulin degludec, or upon crossover from CSII to insulin degludec, the first dose of insulin degludec will be administered on day one and a 50% temporary basal reduction of the insulin pump for 24 hours will be activated. After 24 hours, the insulin pump basal rate will be lowered to the lowest hourly infusion rate (0.025 units per hour or 0.05 units per hour for a total daily basal insulin dose of either 0.6 or 1.2 units per day) for the duration of the insulin degludec treatment arm, with the remainder of the basal insulin dose administered as a single daily Tresiba injection.

The 24 hour basal insulin dose by CSII will be converted to degludec on a unit-for-unit basis. This is because both degludec and CSII are roughly equivalent methods with high efficiency (bioavailability) for delivery of a basal insulin dose. Although there are no head-to-head studies comparing basal insulin dose by CSII to degludec, clinical studies (and the experience of the investigator) suggest that the lowest basal insulin requirement for any given subject will be with either CSII or degludec compared to glargine, NPH or detemir.

A comparison of insulin degludec to continuous subcutaneous infusion of insulin aspart for basal insulin delivery in type 1 diabetes:

#### Visit Procedures

Note: Assessment of hypoglycemia and capturing of AE's (including technical complaints and device site reactions) will be performed at each study visit, as well as diabetes education.

Visit 1 (Screening Visit): Obtain written informed consent; review inclusion/exclusion criteria; demography (including child bearing potential and tobacco use); medical history; record concomitant medications; vital signs (incl. height); complete physical examination; review download of Dexcom and pump; HbA1c, GlycoMark, CBC, comprehensive metabolic profile (CMP), lipid panel, urine microalbumin/creatinine ratio (LabCorp); pregnancy test (urine); review treatment of hypoglycemia; insert Dexcom sensor; provide a hypoglycemia/basal dose diary

Phone Visit 2: Remind subject to insert new Dexcom sensor; assessment of infusion site reactions and occlusions; hypoglycemia assessment (insulin titration if required)

639 640 Visit 3 (Randomization): Review of inclusion/exclusion criteria; vital signs; CGM and insulin 641 pump downloads; HbA1c (POC - Afinion); insulin optimization/titration; dispensing of 642 hypoglycemia/basal dose diary; Tresiba pen teaching (degludec arm only); dispense trial 643 product; treatment questionnaires 644 645 Visit 4: Vital signs; pump and CGM downloads; insulin optimization/titration; assessment of infusion site reactions and occlusions; dispensing of hypoglycemia/basal dose diary 646 647 648 Visit 5: Vital signs; pump and CGM downloads; insulin optimization/titration; assessment of 649 infusion site reactions and occlusions; dispense trial product; dispensing of hypoglycemia/basal 650 dose diary; drug accountability and diabetes education. 651 652 Phone Visit 6: Ensure subject is changing insulin pump sites and CGM per protocol, assessment 653 of infusion site reactions and occlusions; review of hypoglycemia (insulin titration if required) 654 655 Visit 7: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 656 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 657 accountability 658 659 Phone Visit 8: Ensure subject is changing insulin pump sites and CGM per protocol, assessment 660 of infusion site reactions and occlusions; review of hypoglycemia (insulin titration if required) 661 662 Visit 9: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 663 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 664 accountability 665 Visit 10: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 666 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 667 668 accountability 669 670 Visit 11: Dexcom sensor insertion; assessment of infusion site reactions and occlusions, review 671 of hypoglycemia/basal dose diary 672 673 Visit 12 (Cross-over Visit): Vital signs; complete physical examination; pump and CGM 674 downloads; insulin optimization/titration; treatment crossover; Tresiba pen training (degludec 675 arm only); HbA1c, GlycoMark, CBC, comprehensive metabolic profile (CMP), urine microalbumin/creatinine ratio (LabCorp); pregnancy test (urine); dispense trial product; 676 677 treatment questionnaires; dispensing of hypoglycemia/basal dose diary; assessment of infusion 678 site reactions and occlusions; drug accountability 679 680 Visit 13: Vital signs; pump and CGM downloads; insulin optimization/titration; assessment of 681 infusion site reactions and occlusions; dispensing of hypoglycemia/basal dose diary

683 Visit 14: Vital signs; pump and CGM downloads; insulin optimization/titration; assessment of 684 infusion site reactions and occlusions; dispense trial product; dispensing of hypoglycemia/basal 685 dose diary; drug accountability 686 687 Phone Visit 15: Ensure subject is changing insulin pump sites and CGM per protocol, assessment 688 of infusion site reactions and occlusions; review of hypoglycemia (insulin titration if required) 689 690 Visit 16: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 691 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 692 accountability 693 694 Phone Visit 17: Ensure subject is changing insulin pump sites and CGM per protocol, assessment 695 of infusion site reactions and occlusions; review of hypoglycemia (insulin titration if required) 696 697 Visit 18: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 698 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 699 accountability 700 701 Visit 19: Vital signs; pump and CGM downloads; assessment of infusion site reactions and 702 occlusions; dispense trial product; dispensing of hypoglycemia/basal dose diary; drug 703 accountability 704 705 Visit 20: Dexcom sensor insertion; assessment of infusion site reactions and occlusions, review of hypoglycemia/basal dose diary 706 707 708 Visit 21 (End of study visit): Vital signs; complete physical examination; review download of 709 Dexcom and pump; HbA1c, GlycoMark, CBC, comprehensive metabolic profile (CMP), lipid 710 panel, urine microalbumin/creatinine ratio (LabCorp); pregnancy test (urine); review treatment 711 of hypoglycemia; insulin optimization for post-trial treatment; assessment of infusion site 712 reactions and occlusions; drug accountability; treatment questionnaires 713 714 Phone Visit 22 (Follow-up phone visit): Capture AE's; review of hypoglycemia

| Trial Procedures | Screen- | | Random-<br>ization | Treatment Period 1 (First treatment group) | | | | | | | | | | Treatment Period 2 (Second treatment group) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (V), Phone (P) | V1 | P2 | V3 | V4 | V5 | P6 | V7 | P8 | V9 | V10 | V11 | V12 | V13 | V14 | P15 | V16 | P17 | V18 | V19 | V20 | V21 | P22 |
| Timing of Visit (Weeks) | -2 | -1 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 36 | 38 | 40 | 44 |
| Visit Window (Days) | | + 2 | + 1 | + 3 | + 3 | + 3 | + 3 | + 3 | + 3 | + 3 | + 2 | + 3 | + 3 | + 3 | + 3 | + 3 | + 3 | + 3 | + 3 | + 2 | + 3 | + 3 |
| Informed Consent | Х | _ | _ | | _ | _ | _ | _ | _ | _ | _ | | _ | _ | | _ | | _ | | | _ | |
| In/Exclusion Criteria | Х | | Χ | | | | | | | | | | | | | | | | | | | |
| Demography & Tobacco<br>Use | Х | | | | | | | | | | | | | | | | | | | | | |
| Physical Examination | Х | | | | | | | | | | | Х | | | | | | | | | Х | |
| Concomitant Illness | Х | Χ | Х | | | | | | | | | | | | | | | | | | | |
| /Medical History | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant Medication | Χ | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Χ | Χ |
| Child Bearing Potential | Х | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test, Urine | Χ | | | | | | | | | | | Х | | 1 | | | | | | | Х | 1 |
| Height | Χ | | | | | | | | | | | | | | | | | | | | | |
| Body Weight | Χ | | Χ | Х | Х | | Х | | Х | Χ | Χ | Х | Х | Х | | Χ | | Х | Х | Х | Χ | |
| Vital Signs | Χ | | Χ | Х | Х | | Χ | | Χ | Х | Χ | Х | Х | Χ | | Х | | Х | Х | Х | Χ | |
| Dexcom Sensor Insertion | Х | Χ | | | | | | | | | Χ | | | | | | | | | Х | | |
| CGM Download | Х | | Χ | Х | Х | | Х | | Χ | Χ | Χ | Х | Χ | Х | | Х | | Х | Х | Х | Χ | |
| Insulin Pump Download | Χ | | Χ | Х | Х | | Χ | | Χ | Χ | Χ | Х | Χ | Χ | | Χ | | Χ | Х | Х | Χ | |
| Insulin Optimization | | | Χ | Х | Х | | | | | | | Х | Х | Χ | | | | | | | | |
| Blood Sampling | Χ | | Χ | | | | | | | | | Χ | | | | | | | | | Χ | |
| Point-of-Care HbA <sub>1C</sub> | | | Χ | | | | | | | | | | | | | | | | | | | |
| HbA <sub>1C</sub> (central laboratory) | Х | | | | | | | | | | | Х | | | | | | | | | Χ | |
| GlycoMark | Х | | | | | | | | | | | Х | | | | | | | | | Χ | |
| CBC | Х | | | | | | | | | | | Х | | | | | | | | | Χ | |
| CMP | Х | | | | | | | | | | | Х | | | | | | | | | Х | |
| Lipids | Х | | | | | | | | | | | | | | | | | | | | Х | |
| Urine MA | Х | | | | | | | | | | | Х | | | | | | | | | Х | |
| Adverse Events | | | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Hypoglycemia<br>Assessment | X | Х | Х | X | Х | X | X | Х | X | Х | X | X | X | Х | Х | Х | Х | Х | Х | Х | X | Х |
| Technical Complaints | | | | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Infusion Site Reactions | | | | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Х | Χ | Х | Х | Χ | |
| Infusion Site Occlusions | | | | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Χ | Х | Х | Χ | |
| Randomization | | | Х | | | | | | | | | | | | | | | | | | | |
| Dispensing of Trial | | | Χ | | Χ | | Х | | Х | Χ | | Χ | | Х | | Χ | | Х | Х | | | |
| Product | | | | <u></u> | | | | | | | | | | | | | <u> </u> | | | <u> </u> | | <u> </u> |
| Drug Accountability | | | | | Χ | | Χ | | Χ | Χ | | Χ | | Χ | | Χ | | Χ | Χ | | Χ | |
| Treatment Crossover | | | | | | | | | | | | Χ | | | | | | | | | | |
| Questionnaires/Surveys | | | Χ | | | | | | | | | Χ | | | | | | | | | Χ | |
| Diabetes Education | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | |
| REMINDERS | | | | | | | | | | | | | | | | | | | | | | |
| Attend Visit Fasting | X | | | | | | | | | | | Χ | | | | | | | | | Χ | |

| Degludec Pen Instruction | | X* | | | | | | | X* | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Hand out Hypo/Basal | Χ | X | Χ | Χ | Χ | Χ | X | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Dose Diary | | | | | | | | | | | | | | | |

<sup>\*</sup> Dependent upon to which treatment group the subject is assigned.